CLINICAL TRIAL: NCT03806218
Title: Radiofrequency Ablation Using Internally Cooled Wet Electrodes in Bipolar Mode for the Treatment of Recurrent Hepatocellular Carcinoma After Locoregional Treatment: A Randomized Prospective Comparative Study
Brief Title: Bipolar RFA Using Twin ICW Electrodes vs. Switching Monopolar RFA for Recurrent HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNUH-2015-0401
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: RFA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TICW-RFA (Active Comparator): Bipolar RFA using twin internally cooled-wet electrodes
  Interventions: Device: Bipolar RFA; Device: Twin internally cooled-wet electrodes
- SC-RFA (Active Comparator): Switching monopolar RFA using separable clustered electrodes
  Interventions: Device: SM-RFA; Device: Separable clustered electrodes

INTERVENTIONS:
Device: Bipolar RFA — Bipolar RFA in which RF currents flow between two electrodes
  Arms: TICW-RFA
Device: SM-RFA — Monopolar RFA using multiple electrodes with switching mode
  Arms: SC-RFA
Device: Twin internally cooled-wet electrodes — Saline-enhanced twin internally cooled electrodes allow intratumoral injection of a saline solution during the application of the RF current that alters the tissue conductivity
  Other Names: CWTN-T
  Arms: TICW-RFA
Device: Separable clustered electrodes — A separable clustered electrode is similar to a clustered electrode, although it differs from a conventional clustered electrode in that each individual electrode is separable.
  Other Names: Octopus®
  Arms: SC-RFA

SUMMARY:
This study was conducted to provide preliminary data for the main trial to compare efficacy between bipolar radiofrequency ablation (RFA) using twin internally cooled-wet electrodes and switching monopolar RFA using separable clustered electrodes in the treatment of recurrent hepatocellular carcinoma (HCC) after locoregional treatment.

ELIGIBILITY:
Inclusion Criteria:

* radiologic or pathologic diagnosis of HCC recurrence after locoregional treatment
* HCC nodules measuring 1 cm or larger and smaller than 5 cm

Exclusion Criteria:

* more than three HCC nodules
* tumors with major vascular invasion or abutment to the central portal or hepatic vein with a diameter > 5mm
* extrahepatic metastasis
* Child-Pugh class C
* severe coagulopathy (platelet cell count of less than 50,000 cells/mm3 or prothrombin time international normalized ratio (PT-INR) prolongation of more than 50 %)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-05-16 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Minimum diameter of ablation zone per unit time | 3 days after RFA
  Minimum diameter of ablative zone per unit time on post-RFA CT or MRI in a mm.

SECONDARY OUTCOMES:
Technique efficacy | 1 month after RFA
  Technical success on 1 month follow-up imaging after RFA (no residual/progressed tumor)
IDR rate | 12 months, 24 months after RFA
  Cumulative intrahepatic distant recurrence (IDR) rate over 2 years after RFA
EM rate | 12 months, 24 months after RFA
  Cumulative extrahepatic metastasis (EM) rate over 2 years after RFA
Local tumor progression (LTP) | 12 months, 24 months after RFA
  Cumulative LTP rates in two groups in 2 years after RFA

OTHER OUTCOMES:
Complication | 1 month after RFA
  Description and comparison of the type and incidence of major complication after RFA are assessed according to Society of Interventional Radiology (SIR) grading system in two groups.
Volume of ablative zone | 3 days after RFA
  Volume of ablative zone on post-RFA CT or MRI in a mm3
Ablation time | 1 day
  RFA procedure time in each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi JW, Lee JM, Lee DH, Yoon JH, Kim YJ, Lee JH, Yu SJ, Cho EJ. Radiofrequency ablation using internally cooled wet electrodes in bipolar mode for the treatment of recurrent hepatocellular carcinoma after locoregional treatment: A randomized prospective comparative study. PLoS One. 2020 Sep 28;15(9):e0239733. doi: 10.1371/journal.pone.0239733. eCollection 2020. PMID 32986758